CLINICAL TRIAL: NCT01935557
Title: Randomized Comparison of Continuous and Intermittent Heparin Infusion During Catheter Ablation of Atrial Fibrillation
Acronym: COHERE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yong Seog Oh (Other)
Responsible Party: Sponsor-Investigator, Yong Seog Oh, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COHERE
Record Dates: First submitted 2013-09-01; First posted 2013-09-05 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Coagulation; Intravascular
Keywords: Continuous heparin infusion; Intermittent heparin infusion; during catheter ablation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous heparin infusion group (Active Comparator): continuous group is given an initial intravenous heparin 100u/kg and then maintain heparin infusion during procedural.
  Interventions: Drug: Continuous heparin infusion
- Intermittent heparin infusion group (Active Comparator): Intermittent group is given an initial intravenous heparin 100u/kg. Then The ACT is tested every 30min with administration of additional heparin boluses and titration of the heparin drip based on the results and according to the judgment of the operating physician.
  Interventions: Drug: Intermittent heparin infusion

INTERVENTIONS:
Drug: Continuous heparin infusion — continuous group is given an initial intravenous heparin 100u/kg and then maintain heparin infusion during procedural.
  Arms: Continuous heparin infusion group
Drug: Intermittent heparin infusion — Intermittent group is given an initial intravenous heparin 100u/kg. Then The ACT is tested every 30min with administration of additional heparin boluses and titration of the heparin drip based on the results and according to the judgment of the operating physician.
  Arms: Intermittent heparin infusion group

SUMMARY:
Optimal anticoagulation using heparin with close attention to maintain therapeutic dosing during the procedure is important.

Randomized comparison of continuous and intermittent heparin infusion during catheter ablation of Atrial Fibrillation.

DETAILED DESCRIPTION:
Intravenous heparin was used during the procedure to prevent catheter-induced thrombosis.

heparin is administered during the procedure to achieve recommended activation clotting times (ACT) values, typically >300 seconds to prevent thromboemboli during the procedure.

Most of the practitioners was that ACT level should be checked at 30- to 60-minute intervals and then have injected intermittently.

intermittent heparin infusion, concentration is great changed because the heparin has 30minutes half-period.

researchers postulate that a constant therapeutic concentrations would be beneficial to continuous infusion than intermittent infusion.

ELIGIBILITY:
Inclusion Criteria:

* Atrial Fibrillation, Radiofrequency catheter ablation scheduled

Exclusion Criteria:

* Clinical trial denied

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2012-12; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
therapeutic ACT retention rate during procedure | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yong Seog Oh, MD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul st. mary's hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim TS, Kim SH, Kim BK, Kim JY, Kim JH, Jang SW, Lee MY, Rho TH, Oh YS. Randomized Comparison of Continuous Versus Intermittent Heparin Infusion During Catheter Ablation of Atrial Fibrillation. JACC Clin Electrophysiol. 2016 Jun;2(3):319-326. doi: 10.1016/j.jacep.2015.11.004. Epub 2015 Dec 9. PMID 29766891